CLINICAL TRIAL: NCT04557852
Title: Clinical Outcome and Urodynamic Changes of Tailored Transvaginal Mesh Surgery for Pelvic Organ Prolapse: a Mid-term Follow-up With a Median Duration of 30 Months
Brief Title: Mid-term Follow-up for Tailored ATVM
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202006093RIND
Record Dates: First submitted 2020-09-08; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-07

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Pelvic organ prolapse; Transvaginal mesh; lower urinary tract symptoms; Urodynamic study
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anterior transvaginal mesh group: Women received anterior transvaginal mesh surgery without concomitant mid-urethral sling surgery.
  Interventions: Procedure: ATVM

INTERVENTIONS:
Procedure: ATVM — Tailored anterior transvaginal mesh for pelvic organ prolapse

SUMMARY:
Lower urinary tract symptoms may change after pelvic organ prolapse surgery. Thus, the aim of this study was to elucidate (1) the changes of lower urinary tract symptoms and (2) the changes in values of urodynamic parameters between baseline and after pelvic organ prolapse surgery.

DETAILED DESCRIPTION:
Between November 2011 and December 2015, medical records of all consecutive women who underwent anterior transvaginal mesh surgery (ATVM) but without concomitant mid-urethral sling surgery were reviewed. Data of pre- and post-operative lower urinary tract symptoms and urodynamic parameters were compared. The bladder outlet obstruction was defined when the detrusor pressure at maximum flow rate was not less than 40cmH2O, and the maximum flow rate was less than 12 mL/s. Overactive bladder syndrome, detrusor overactivity, bladder oversensitivity and urodynamic stress incontinence were also recognized as international continence society definition. STATA software was used for statistical analysis. Wilcoxon signed-rank test or McNemar's test was used for statistical analysis as appropriate. P < 0.05 was considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Women with pelvic organ prolapse
* Women received anterior transvaginal mesh surgery

Exclusion Criteria:

* Concomitant mid-urethral sling surgery
* Chronic urinary tract infection
* Interstitial cystitis
* Malignancy history in pelvic organ
* Ever received pelvic radiation
* Concomitant transabdominal surgery

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between November 2011 and December 2015, medical records of all consecutive women who underwent anterior transvaginal mesh surgery for their advanced pelvic organ prolapse were reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Voiding difficulty | November 2011 to December 2015
  Weak stream of urination, intermittency, strain to void or incomplete empty sensation after the anterior transvaginal mesh surgery

SECONDARY OUTCOMES:
Overactive bladder syndrome | November 2011 to December 2015
  Urinary urgency, with or without incontinence, may accompany with urinary frequency and nocturia.

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD will be shared under reasonable request

REFERENCES:
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Result] Wu PC, Wu CH, Lin KL, Liu Y, Loo Z, Lee YC, Long CY. Predictors for de novo stress urinary incontinence following pelvic reconstruction surgery with transvaginal single-incisional mesh. Sci Rep. 2019 Dec 16;9(1):19166. doi: 10.1038/s41598-019-55512-0. PMID 31844157
- [Result] Long CY, Wang CL, Lin KL, Ker CR, Loo Z, Liu Y, Wu PC. Laparoscopic Long Mesh Surgery with Augmented Round Ligaments: A Novel Uterine Preservation Procedure For Apical Pelvic Organ Prolapse. Sci Rep. 2020 Apr 20;10(1):6615. doi: 10.1038/s41598-020-63725-x. PMID 32313187
- [Result] Chang TC, Hsiao SM, Chen CH, Wu WY, Lin HH. Clinical Outcomes and Urodynamic Effects of Tailored Transvaginal Mesh Surgery for Pelvic Organ Prolapse. Biomed Res Int. 2015;2015:191258. doi: 10.1155/2015/191258. Epub 2015 Nov 8. PMID 26634203
- [Result] Chang TC, Hsiao SM, Wu PC, Chen CH, Wu WY, Lin HH. Comparison of clinical outcomes between tailored transvaginal mesh surgery and native tissue repair for pelvic organ prolapse. J Formos Med Assoc. 2019 Dec;118(12):1623-1632. doi: 10.1016/j.jfma.2019.08.034. Epub 2019 Sep 18. PMID 31542332